CLINICAL TRIAL: NCT01193192
Title: A Retrospective Analysis of Neevo® and NeevoDHA® Compared to a Standard Prenatal Vitamin in Anemia During Pregnancy
Status: Terminated | Type: Observational
Why Stopped: Inadequate number of charts available for Test Group
Sponsor: Pamlab, L.L.C. (Industry)
Collaborators: Baylor Health Care System (Other); Norman Regional Health System (Unknown); Five Oaks Medical Group (Unknown)
Responsible Party: Sponsor
Organization: Pamlab, Inc. (Industry)
Other Study IDs: N-002
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Anemia in Pregnancy; Pre-eclampsia
Keywords: Neevo; Neevo DHA; L-methylfolate; anemia during pregnancy; folic acid; vitamin B12; prenatal vitamins; hemoglobin; iron deficiency; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Iron Deficiencies | interventions — Prenatal Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm #1 (Test Group): 100 subject administered Neevo® or NeevoDHA® daily
  Interventions: Other: Neevo®
- Arm #2 (Control group): 100 subject administered a prenatal vitamin daily
  Interventions: Other: Prenatal vitamins

INTERVENTIONS:
Other: Neevo® — A prenatal "medical food" - analogous to a prenatal vitamin but containing L-methylfolate in addition to folic acid
  Groups: Arm #1 (Test Group)
Other: Prenatal vitamins — for inclusion in the Control Group, prenatal vitamins must have contained ≤1mg folic acid, 27 - 35mg iron, and ≤12mcg vitamin B12.
  Groups: Arm #2 (Control group)

SUMMARY:
This study is a multi-site, retrospective chart review to determine the effect of Neevo® or NeevoDHA® (with higher folate and B12) versus standard prenatal vitamins on hemoglobin (Hgb) levels in pregnant women throughout the course of pregnancy. Neevo® is a prescription medical food indicated for the dietary management of women under a doctor's care who face high risk pregnancies, older overactive bladder (OB) patients and patients unable to fully metabolize folic acid. Data will be collected from existing patient charts of subjects administered Neevo® or NeevoDHA® daily compared to subjects administered a prenatal vitamin daily.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females, age 21-39, who received either Neevo®/NeevoDHA® or another standard prenatal vitamin (Prenatal vitamins must contain ≤1 mg folic acid, 27-35mg iron, and ≤12mcg vitamin B12).
* Clinical diagnosis of pregnancy must have been made at ≤12 weeks of Pregnancy, and delivery must have occurred on or after January 1, 2008 and on or before March 31, 2010
* Subjects must have been compliant in taking Neevo®/NeevoDHA® or other prenatal vitamin

Exclusion Criteria:

* Subjects should not have taken Prenate®, Prenate®DHA, or Prenate® Elite, which are L-methylfolate-containing prenatal vitamins.
* The following supplements within 2 months of diagnosis of pregnancy: B12 injection; > 35mg Iron; > 1.2 mg of folate; or a L-methylfolate product that is not a prenatal vitamin such as Life Extension methylfolate, Prothera methylfolate, Thorne 5-MTHF, Metanx®, Deplin®, Cerefolin®, or CerefolinNAC®
* History of leukemia or any anemia other than iron deficiency anemia or;
* Taking any iron supplement (in addition to the prenatal vitamin) prior to Week 22

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women Who Received Neevo®/NeevoDHA® or Another Standard Prenatal Vitamin
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Mean Hemoglobin (Hgb) Levels | At the time of diagnosis of pregnancy, at the end of the second trimester (Weeks 22-28), and at delivery.
  To determine the effect of Neevo®/NeevoDHA® versus standard prenatal vitamins on mean hemoglobin (Hgb) levels in pregnant women throughout the course of pregnancy.

SECONDARY OUTCOMES:
Mean Change in Hemoglobin (Hgb) Levels | At the time of diagnosis of pregnancy, at the end of the second trimester (Weeks 22-28), and at delivery.
  To determine the effect of Neevo®/NeevoDHA® versus standard prenatal vitamins on mean change in hemoglobin levels in pregnant women.
Incidence of Anemia | At the time of diagnosis of pregnancy, at the end of the second trimester (Weeks 22-28), and at delivery.
  To determine if Neevo®/NeevoDHA® administration during pregnancy results in fewer incidences of anemia than with standard prenatal vitamins.
Incidence of Pre-eclampsia | At the time of diagnosis of pregnancy, at the end of the second trimester (Weeks 22-28), and at delivery.
  To determine if Neevo®/NeevoDHA® administration during pregnancy results in fewer cases of pre-eclampsia than with standard prenatal vitamins.
Mean Infant Birth Rate | At the time of diagnosis of pregnancy, at the end of the second trimester (Weeks 22-28), and at delivery.
  To determine the effect of Neevo®/NeevoDHA® versus standard prenatal vitamins on infant birth weight.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Jarvis, M.D., Principal Investigator — Norman Regional Health System
Locations (2):
- United States (2):
  - Five Oaks Medical Group, Chickasha, Oklahoma
  - Norman Regional Health System, Norman, Oklahoma

REFERENCES:
- [Derived] Bentley S, Hermes A, Phillips D, Daoud YA, Hanna S. Comparative effectiveness of a prenatal medical food to prenatal vitamins on hemoglobin levels and adverse outcomes: a retrospective analysis. Clin Ther. 2011 Feb;33(2):204-10. doi: 10.1016/j.clinthera.2011.02.010. Epub 2011 Mar 25. PMID 21440300